CLINICAL TRIAL: NCT06664736
Title: Effects of Home-Based Exercise Program in Children After Acute Lymphoblastic Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ilke Keser, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 419 Haspolat M
Record Dates: First submitted 2024-10-20; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-09

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: leukemia; acute lymphoblastic; interleukins; inflammation; exercise
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Inflammation; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise (Experimental): The exercise group performed a home-based exercise program consisting of aerobics 3 days a week and strengthening and stretching exercises 2 days a week, with videos and infographics, for 8 weeks.
  Interventions: Behavioral: Exercise
- Control (Other): control group was advised to increase physical activity.
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Exercise — The exercise group performed a home-based exercise program consisting of aerobics 3 days a week with videos and strengthening and stretching exercises 2 days a week with infographics, for 8 weeks.
  Arms: Exercise
Behavioral: Physical activity — The control group was advised to increase physical activity
  Arms: Control

SUMMARY:
This prospective randomized controlled study aimed to investigate the effects of a home-based exercise program on physical functions, inflammatory markers, and Brain-Derived Neurotrophic Factor (BDNF) in children followed after Acute Lymphoblastic Leukemia (ALL) treatments. Ankle dorsiflexion range of motion (ROM), dorsiflexion and knee extensor muscle strength, hand grip strength, aerobic endurance, and functional mobility were assessed using a goniometer, digital dynamometer; hand dynamometer, 6 Minute Walk Test (6 MWT), Timed Up and Go Test respectively. Interleukin-1 Beta, Tumor Necrosis Factor-Alpha, Interleukin-6 (IL-6), and BDNF values were examined using ELISA kits. 20 patients will be included in the study. The patients randomly divided into 2 groups: exercise (n:10) and control (n:10). The exercise group performed a home-based exercise program consisting of aerobics 3 days a week and strengthening and stretching exercises 2 days a week, with videos and infographics, for 8 weeks. The control group was advised to increase physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 6-18,
* Having clinical diagnose of Acute Lymphoblastic Leukemia,
* Being completed medical treatment

Exclusion Criteria:

* Having a history of neurological, developmental, or genetic disorders,
* Communicating problems
* Medical conditions such as advanced cardiac damage, decreased bone quality, acute infection, and cancer recurrence.

Children who could not accomplish the exercises and evaluations, who did not want to continue the study, who could not be contacted for more than 2 weeks, and who disrupted the exercise program for more than 2 weeks were excluded from the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Difference between baseline and final active ankle dorsiflexion range of motion | 8 weeks
  Active ankle dorsiflexion ROM was evaluated with a Baseline® (Aurora, IL, USA) brand goniometer in a supine position, with the knee supported by a pillow and the knee flexed and recorded in degrees
Difference between baseline and final muscle strength | 8 weeks
  Knee extensor and ankle dorsiflexor muscle strength were assessed using a digital handheld dynamometer (Lafayette Instrument Company, Lafayette, Indiana). The "break" technique was used to measure muscle strength.
Difference between baseline and final handgrip strength | 8 weeks
  Handgrip strength was evaluated using a hand dynamometer (J-Tech Commander Grip Track Dynamometer, JTECH Medical, Midvale, UT, US).The patient was positioned in a sitting position with the shoulder adducted and neutrally rotated, the elbow at 90° flexion, and the forearm and wrist in neutral. The patient was asked to squeeze the device as hard as he could for 5 seconds, and during the measurement, the child was given verbal encouragement such as "squeeze as hard as you can." Measurements were repeated 3 times and the average value was recorded in Newtons.
Difference between baseline and final aerobic endurance | 8 weeks
  Aerobic endurance was evaluated using the 6-minute walk test (6MWT). 6MWT was performed by the American Thoracic Society guidelines. During the test, the patient was asked to walk in the corridor as fast as he could without running, jumping, or jumping within the determined limits for 6 minutes. Total walking distance was recorded in meters
Difference between baseline and final functional mobility | 8 weeks
  Functional mobility was assessed with the Timed Up and Go Test. While the patient was in a sitting position on an armless chair, he was asked to get up on command, walk 3 meters, return, and sit on the chair again. The elapsed time was recorded in seconds.
Difference between baseline and final serum inflammatory markers and brain derived neurotrophic factor levels | 8 weeks
  Serum samples required to examine levels of inflammatory markers (IL-6, TNF-a, and IL-1b) and BDNF were obtained during blood collection at the patients' routine hospital visits.Data about serum IL-6 and TNF-a were recorded from the hospital information system. Serum IL-1b and BDNF levels were analyzed using ELISA kits provided by the researchers.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No